CLINICAL TRIAL: NCT03647657
Title: 177Lu-PP-F11N in Combination With Sacubitril for Receptor Targeted Therapy and Imaging of Metastatic Thyroid Cancer (Lumed Phase 0/B)
Brief Title: 177Lu-PP-F11N in Combination With Sacubitril for Receptor Targeted Therapy and Imaging of Metastatic Thyroid Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other); Center for Proton Therapy, Paul Scherrer Institute, Villigen,Switzerland (Other); University Hospital, Zürich (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-00972
Record Dates: First submitted 2018-08-20; First posted 2018-08-27 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Thyroid Cancer, Medullary
Keywords: Calcitonin; Medullary thyroid carcinoma; Peptide receptor radionuclide therapy; Gastrin; Cholecystokinin-2 receptor
MeSH Terms: conditions — Thyroid cancer, medullary; Carcinoma, Medullary | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Intervention Model Description: Group 1 patients will receive first 177Lu-PP-F11N alone, second 177Lu-PP-F11N in combination with Sacuitril. Group 2 patients will first receive 177Lu-PP-F11N in combination with Sacuitril, second 177Lu-PP-F11N alone. Affiliation of patients to Groups 1 and 2 will be randomised.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entresto second (Experimental): First intravenous application of 2 x 1 gigabequerel (GBq) 177Lu-PP-F11N without and second injection with additional medication of Sacuitril (100 mg Entresto)(crossover)
  Interventions: Drug: 177Lu-PP-F11N; Drug: Sacuitril
- Entresto first (Experimental): First intravenous application of 2 x 1 gigabequerel (GBq) 177Lu-PP-F11N with and second injection without additional medication of Sacuitril (100 mg Entresto)(crossover)
  Interventions: Drug: 177Lu-PP-F11N; Drug: Sacuitril

INTERVENTIONS:
Drug: 177Lu-PP-F11N — Intravenous application of 2 x 1 gigabequerel (GBq) 177Lu-PP-F11N with and without co-medication with Sacuitril (100 mg Entresto) in each patient
  Other Names: Radiopharmakon
Drug: Sacuitril — Medication with Sacuitril (100 mg Entresto) additional to the injection of 177Lu-PP-F11N
  Other Names: Entresto

SUMMARY:
The purpose of this study is to determine the use of 177Lu-PP-F11N for imaging and therapy of patients with advanced medullary thyroid carcinoma (MTC). 177Lu-PP-F11N is a gastrin analogon, binding to cholecystokinin-2 receptors. This receptors show an overexpression on more than 90 % of medullary thyroid carcinomas.

DETAILED DESCRIPTION:
A phase 0 study (Lumed study part A) was already performed, showing low toxicity of 177Lu-PP-F11N and tumor uptake in all patients. Co-injection of Physiogel (Gelofusin) showed insignificant reduction of kidney uptake and can therefore be omitted for a radionuclide therapy with 177Lu-PP-F11N. In this study, the effect of the NEP-1 inhibitor Sacuitril on the in-vivo stability of 177Lu-PP-F11N and the uptake, respectively radiation doses in MTC metastases and organs will be evaluated, using a cross-over design already used for the Lumed part A study. Each patient will receive two injections of 177Lu-PP-F11N, with and without additional medication with Sacuitril Imaging findings, acquired by SPECT/CT, will be compared to imaging with 68Ga-DOTATOC positron emission tomography (PET)/CT. The inclusion of 8 patients is planned.

ELIGIBILITY:
Inclusion Criteria:

* Advanced MTC with elevated levels of calcitonin (> 100 pg/ml) and/or calcitonin-doubling time < 24 months before or after total thyroidectomy
* 68Ga-DOTATOC PET/CT not older than 12 weeks
* Age > 18 years
* Informed consent

Exclusion Criteria:

* Medication with Vandetanib 3 weeks before the study and during the study
* Renal failure (calculated glomerular filtration rate (GFR) < 60 ml/min per 1.73 m2 body surface).
* Bone marrow failure (thrombocytes < 70 000/μl, leucocytes < 2 500/μl, hemoglobin < 8 g/dl).
* Pregnancy and breast feeding
* Known, serious side reaction in the case of a former application of pentagastrin
* Active, second malignancy oder remission after second malignancy < 5 years
* Age over 64 years
* Systolic bood pressure < 112 mmHg at the time of screening
* Simultaneous medication with angiotensin converting enzyme (ACE)-inhibitors, or withdrawal for less than 36 h prior to the medication with Entresto or simultaneous medication with AT-II-receptor blockers
* Known intolerance to Sacubitril or Valsartan
* Known angioedema in anamnesis in the context of a medication with an ACE-inhibitor or an AT-II-receptor blocker

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Tumor radiation doses | Measurement up to 72 hours after each injection of 177Lu-PP-F11N
  Evaluation of the radiation doses in tumor tissue from MTC after injection of 177Lu-PP-F11N alone and in combination with Sacuitril (Entresto)

SECONDARY OUTCOMES:
Kidney radiation doses | Measurement up to 72 hours after each injection of 177Lu-PP-F11N
  Evaluation of the radiation doses in the kidneys and the tumor-to-kidney dose ratios after injection of 177Lu-PP-F11N alone and in combination with Sacuitril (Entresto)
Organ radiation doses | Measurement up to 72 hours after each injection of 177Lu-PP-F11N
  Evaluation of the radiation doses in other organs and the appropriate organ-to-kidney dose ratios after injection of 177Lu-PP-F11N alone and in combination with Sacuitril (Entresto)
In-vivo stability | Blood samples for measurement 5 and 30 minutes post injection of 177Lu-PP-F11N
  Measurement (HPLC) of the in-vivo stability of 177Lu-PP-F11N alone and in combination with Sacuitril (Entresto).
Autoradiography | Through study completion, up to 18 months
  In case of surgery with available tumor tissue samples, imaging results will be compared with autoradiographic analysis of somatostatine- and CCK2-receptor expression in tumor tissue.

OTHER OUTCOMES:
Chromogranin A | Measurement up to 72 hours after the first injection of 177Lu-PP-F11N
  Chromogranin A blood values will be compared to the radiation doses of the stomach.
68Ga-DOTATOC PET/CT | Measurement up to 72 hours after each injection of 177Lu-PP-F11N
  Comparison of tumor imaging by 68Ga-DOTATOC PET/CT and 177Lu-PP-F11N SPECT/CT

CONTACTS AND LOCATIONS:
Overall Officials: Christof Rottenburger, Dr. med., Principal Investigator — University Hospital Basel, Clinic for radiology and nuclear medicine; Damian Wild, PhD Dr, Study Director — University Hospital Basel, Clinic for radiology and nuclear medicine
Locations (1):
- University Hospital Basel, Clinic for radiology and nuclear medicine, Basel, Switzerland

REFERENCES:
- [Result] Sauter AW, Mansi R, Hassiepen U, Muller L, Panigada T, Wiehr S, Wild AM, Geistlich S, Behe M, Rottenburger C, Wild D, Fani M. Targeting of the Cholecystokinin-2 Receptor with the Minigastrin Analog 177Lu-DOTA-PP-F11N: Does the Use of Protease Inhibitors Further Improve In Vivo Distribution? J Nucl Med. 2019 Mar;60(3):393-399. doi: 10.2967/jnumed.118.207845. Epub 2018 Jul 12. PMID 30002107
- [Derived] Rottenburger C, Hentschel M, Furstner M, McDougall L, Kottoros D, Kaul F, Mansi R, Fani M, Vija AH, Schibli R, Geistlich S, Behe M, Christ ER, Wild D. In-vivo inhibition of neutral endopeptidase 1 results in higher absorbed tumor doses of [177Lu]Lu-PP-F11N in humans: the lumed phase 0b study. EJNMMI Res. 2024 Apr 6;14(1):37. doi: 10.1186/s13550-024-01101-w. PMID 38581480
- See also: University Hospital Basel Homepage — https://www.unispital-basel.ch/en